CLINICAL TRIAL: NCT06060275
Title: Neurofilament Light Chain as a Potential Marker in Behcet's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nayera Ahmed Abdelhamed, Nayera Ahmed Abdelhamed, Assiut University
Other Study IDs: Neurofilament in behcet
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Behçet
MeSH Terms: conditions — Behcet Syndrome | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum sample and nerve conduction study and cerebrospinal fluid study — serum sample and cerebrospinal fluid study to detect Neurofilament light chain Nerve conduction study

SUMMARY:
To determine the role of neurofilament light chain in Behçet's disease with or without neurological affection and its relation to neurological manifestation (either peripheral or central ).

DETAILED DESCRIPTION:
Behçet disease is a multisystemic autoinflammatory disorder characterized by recurrent oral and genital ulcer, eye affection, thrombosis and many systems can be affected with the most serious being the nervous system affection which is commonly called neuro-Behçet's disease (NBD) In Ghita et al, the prevalence of Behcet disease in Egypt was estimated to be 3.6/100,000 with CNS affection occurred in about 13.1% of the patients , while in other study performed in Egypt the peripheral neuropathy affection reached 53.3% of the patients with insignificant difference between both upper and lower limb but sensory affection was manifested more than motor affection in those patients.

Neurofilament light chain (NFL) is a neuronal cytoplasmic protein, which was assumed to have a role as a prognostic biomarker in several neuroimmunological and neurodegenerative diseases. It was documented in peripheral nerve affection of patients with diabetes mellitus and GuillainBarré syndrome. Recently, some studies documented the presence of high level of NFL chain in serum of neurolupus and primary sjogren's diseases , more over in 2022, Karaaslan et al. measured NFL in the cerebrospinal fluid (CSF) and found it high in neurobehcet patients and assumed that it can predict the prospective cognitive and somatic disability in NBD patients.

So, the investigators aim at our study to assess the role of NFL chain in serum of behcet disease in those with and without peripheral and central nervous system affection and its relation to neurological manifestation.

ELIGIBILITY:
Inclusion Criteria:

* any adult patient satisfied International study group criteria of Behcet's disease

Exclusion Criteria:

* Patients with definite diagnosis for any other causes affecting central and peripheral nervous system eg….

  1. Infection (Viral, Bacterial, Fungal)
  2. Toxic
  3. Drug induced
  4. Other diseases (Multiple sclerosis, Neuromyelitis Optica)
  5. Trauma
  6. other autoimmune diseases
  7. Diabetic patients
  8. purely degenerative diseases
  9. Tumours

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - any adult patient satisfied International study group criteria of Behcet's disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
aim at our study to assess the role of NFL chain in serum of behcet disease in those with and without peripheral and central nervous system affection and its relation to neurological manifestation | baseline
  compare the level of NFL in serum between groups of Behcet patients with or without central and peripheral Nervous system affection

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Makarem, Study Director — Assiut University; Rania Gamal, Principal Investigator — Assiut University

REFERENCES:
- [Background] Davatchi F, Chams-Davatchi C, Shams H, Shahram F, Nadji A, Akhlaghi M, Faezi T, Ghodsi Z, Sadeghi Abdollahi B, Ashofteh F, Mohtasham N, Kavosi H, Masoumi M. Behcet's disease: epidemiology, clinical manifestations, and diagnosis. Expert Rev Clin Immunol. 2017 Jan;13(1):57-65. doi: 10.1080/1744666X.2016.1205486. Epub 2016 Jul 11. PMID 27351485
- [Background] Gheita TA, El-Latif EA, El-Gazzar II, Samy N, Hammam N, Abdel Noor RA, El-Shebeiny E, El-Najjar AR, Eesa NN, Salem MN, Ibrahim SE, El-Essawi DF, Elsaman AM, Fathi HM, Sallam RA, El-Shereef RR, Abd-Elazeem MI, Said EA, Khalil NM, Shahin D, El-Saadany HM, ElKhalifa MS, Nasef SI, Abdalla AM, Noshy N, Fawzy RM, Saad E, Moshrif AH, El-Shanawany AT, Abdel-Fattah YH, Khalil HM; Egyptian College of Rheumatology-Behcet's Disease Study Group (ECR-BDSG). Behcet's disease in Egypt: a multicenter nationwide study on 1526 adult patients and review of the literature. Clin Rheumatol. 2019 Sep;38(9):2565-2575. doi: 10.1007/s10067-019-04570-w. Epub 2019 May 22. PMID 31119493
- [Background] Karaaslan Z, Sanli E, Timirci-Kahraman O, Yilmaz V, Akbayir E, Koral G, Icoz S, Gunduz T, Kucukali CI, Kurtunvu M, Tuzun E. Cerebrospinal fluid level of neurofilament light chain is associated with increased disease activity in neuro-Behcet's disease. Turk J Med Sci. 2022 Aug;52(4):1266-1273. doi: 10.55730/1300-0144.5432. Epub 2022 Aug 10. PMID 36326394
- [Background] Maalmi H, Strom A, Petrera A, Hauck SM, Strassburger K, Kuss O, Zaharia OP, Bonhof GJ, Rathmann W, Trenkamp S, Burkart V, Szendroedi J, Ziegler D, Roden M, Herder C; GDS Group. Serum neurofilament light chain: a novel biomarker for early diabetic sensorimotor polyneuropathy. Diabetologia. 2023 Mar;66(3):579-589. doi: 10.1007/s00125-022-05846-8. Epub 2022 Dec 6. PMID 36472640
- [Background] Engel S, Boedecker S, Marczynski P, Bittner S, Steffen F, Weinmann A, Schwarting A, Zipp F, Weinmann-Menke J, Luessi F. Association of serum neurofilament light chain levels and neuropsychiatric manifestations in systemic lupus erythematosus. Ther Adv Neurol Disord. 2021 Oct 22;14:17562864211051497. doi: 10.1177/17562864211051497. eCollection 2021. PMID 34707690
- [Background] Tjensvoll AB, Lauvsnes MB, Zetterberg H, Kvaloy JT, Kvivik I, Maroni SS, Greve OJ, Beyer MK, Hirohata S, Putterman C, Alves G, Harboe E, Blennow K, Goransson LG, Omdal R. Neurofilament light is a biomarker of brain involvement in lupus and primary Sjogren's syndrome. J Neurol. 2021 Apr;268(4):1385-1394. doi: 10.1007/s00415-020-10290-y. Epub 2020 Oct 30. PMID 33128084